CLINICAL TRIAL: NCT01407536
Title: Effect of Thermal Stimulation on Cortical Excitability and Motor Function in Chronic Stroke Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other); Kaohsiung Medical University (Other)
Responsible Party: Jau-Hong Lin/Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSC-96-2314-B-037-028-MY3
Record Dates: First submitted 2011-06-26; First posted 2011-08-02 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-06

CONDITIONS: Stroke
Keywords: Stroke; Thermal Stimulation; Upper Extremity; Motor Recovery; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Thermal stimulation system — The subjects meeting our criteria will be randomly assigned to either the experimental group (EXP) or the control group (COT). The EXP and COT received upper extremity thermal stimulation protocol for 30 minutes a day for 20 days. The TS temperature of EXP for noxious stimulation was set at 46-47°C for heat and 7-8°C for cold stimulation; the temperature of COT for innoxious stimulation was set at 40°C for warm and 20°C for cold stimulation.

SUMMARY:
Functional magnetic resonance imaging (fMRI) has confirmed that thermal stimulation (TS) may facilitate cortical excitability in healthy adults. However, it is unknown whether TS can increase cortical excitability in stroke patients. Compared to the fMRI, the transcranial magnetic stimulation (TMS) possesses more concise conditions in temporal resolution, and it can present the cerebrum activation situation more instantaneously. This study aimed to use TMS examining the effect on corticomotor excitability, reorganization and functional motor recovery after TS on affected upper limbs of chronic stroke patients.

DETAILED DESCRIPTION:
The study was an assessor-blinded randomized controlled clinical trial. The participants (more than 3 months posts-stroke)were randomly assigned to experiment (EXP) and control (COT) groups. All participants received regular conventional rehabilitation programs. The EXP and COT received additional upper extremity TS protocol for 30 minutes a day for 20 days. The TS temperature of EXP for noxious stimulation was set at 46-47°C for heat and 7-8°C for cold stimulation; the temperature of COT for innoxious stimulation was set at 40°C for warm and 20°C for cold stimulation. The motor and sensory performance were evaluated at baseline and post-20th- TS by Brunnstrom's recovery stage, Modified Ashworth Scale (MAS), Barthel Index (BI), Upper Extremity Subscale of the Fugl-Meyer Motor Function Assessment (UE-FM) and Thermal Quantitative Sensory Testing (tQST). At pre-1st-TS, post-1st-TS, post-10th-TS and post-20th-TS, focal TMS was used to obtain measurement of motor threshold (MT), motor evoked potentials (MEPs), size of cortical motor output map and location of the amplitude-weighted centre of gravity of the motor output map (CoG) from abductor pollicis brevis (APB) in bilateral upper extremities.

ELIGIBILITY:
Inclusion Criteria:

1. first-ever stroke survivors with unilateral hemispheric lesions from a ischemic stroke.
2. stroke onset more than 3 months
3. no severe cognitive impairments and able to follow instructions
4. the ability to sit on a chair for more than 30 minutes independently
5. no family history of epilepsy

Exclusion Criteria:

1. musculoskeletal or cardiac disorders that could potentially interfere with experimental tests;
2. diabetic history or sensory impairment attributable to peripheral vascular disease or neuropathy;
3. speech disorder or global aphasia;
4. participating in any experimental rehabilitation or drug studies;
5. skin injuries, burns, or fresh scars at the sites of stimulation;
6. contraindication of heat or ice application

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Transcranial Magnetic Stimulation | Change from baseline in cortical excitability at post-1st-intervention, post-10th-intervention, post-20th-intervention and 1 month follow-up

SECONDARY OUTCOMES:
Modified Ashworth Scale | baseline, post-20th-intervention, 1 month follow-up
Barthel Index | baseline, post-20th-intervention, 1 month follow-up
Upper Extremity Subscale of the Fugl-Meyer Motor Function Assessment | baseline, post-20th-intervention, 1 month follow-up
Thermal Quantitative Sensory Testing | baseline, post-20th-intervention, 1 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jau Hong Lin, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Department of Physical Therapy, Kaohsiung Medical University, Kaohsiung, Taiwan, Kaohsiung City, Taiwan